CLINICAL TRIAL: NCT04583592
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy of Camostat Mesilate for Treatment of COVID-19 in Outpatients
Brief Title: Camostat Efficacy vs. Placebo for Outpatient Treatment of COVID-19 (CAMELOT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sagent Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NI03-CV19-001
Record Dates: First submitted 2020-10-07; First posted 2020-10-12 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Camostat Mesilate (Experimental): Participants will receive camostat mesilate for 14 days in addition to standard of care treatment.
  Interventions: Drug: Camostat Mesilate
- Placebo (Placebo Comparator): Participants will receive placebo for 14 days in addition to standard of care treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Camostat Mesilate — Camostat mesilate administered as oral 100 mg round tablets. Study dose: Two 100 mg tablets (200 mg total) taken orally 4 times daily for 14 days.
  Other Names: Camostat Mesylate; Foipan®
  Arms: Camostat Mesilate
Drug: Placebo — Placebo administered as oral round tablets. Study dose: Two placebo tablets taken orally 4 times daily for 14 days.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of camostat mesilate in ambulatory patients with confirmed COVID-19 with at least one risk factor for severe illness.

DETAILED DESCRIPTION:
Participants will be randomized in a 2:1 ratio of camostat:placebo. Approximately 300 participants are planned to be enrolled (200 participants to camostat mesilate and 100 participants to placebo). Participants will be treated with camostat mesilate 200 mg or placebo drug orally 4 times a day for 14 days, and receive local standard of care (SOC) in addition to study drug. Participants will be followed until Day 28. Participants will be seen in the clinic for assessments, blood draws, and mid-turbinate nasal samples on Screening/Day 1, Day 7, Day 15 and early termination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults willing and able to provide informed consent before performing study procedures
2. Adults ≥18 years of age at time of informed consent
3. Participants must have written notification of laboratory confirmed COVID-19 infection performed prior to screening, at a local laboratory by RT-PCR or other commercial or public health assay in any specimen; and participants must be randomized within 72 hours of receiving the above notification of laboratory confirmed COVID-19
4. Have a mild or moderate form of COVID-19 defined as SpO2 > 94% at screening
5. Participants must have at least 1 of the following risk factors for severe illness

   1. Aged 65 years or older
   2. Hypertension
   3. Diabetes mellitus
   4. Chronic lung disease including asthma, chronic obstructive pulmonary disease (COPD), and interstitial lung disease (eg, idiopathic pulmonary fibrosis)
   5. Chronic cardiac conditions, including coronary artery disease (CAD), heart failure, congenital heart disease, cardiomyopathy
   6. Severe obesity (body mass index [BMI] ≥ 40 kg/m^2)
   7. Chronic liver disease, including cirrhosis
6. Must agree not to enroll in another study of an investigational agent or take any other drug that has been granted Emergency Use Authorization prior to completion of Day 28
7. If women of childbearing potential (WOCBP) or men whose sexual partners are WOCBP, must be able and willing to use at least 1 highly effective method of contraception during the study and for 90 days after receiving the last dose of study drug

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in participants' best interest, or has any condition that does not allow the protocol to be followed safely
2. Known severe liver disease (eg, Child Pugh score > 12, AST >5 times upper limit)
3. SaO2/SPO2 ≤94% on room air condition, or the Pa02/Fi02 ratio < 300 mgHg
4. Known allergic reaction to camostat mesilate or one of its excipients
5. Known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m^2) or receiving dialysis
6. Pregnant or breastfeeding, or positive pregnancy test in a predose examination
7. Receipt of any experimental treatment for COVID-19, including agents with demonstrated or possible direct acting antiviral activity, including, but not limited to, remdesivir, hydroxychloroquine, lopinavir/ritonavir, tocilizumab, or ivermectin, within the 30 days prior to the time of the screening evaluation. No off label use of a drug for COVID 19 is allowed.
8. History of human immunodeficiency virus infection on highly active antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Palmtree Clinical Research, Inc. (Site 125), Palm Springs, California
  - Synergy Healthcare, LLC (Site 124), Bradenton, Florida
  - Clinical Research of Brandon, LLC (Site 123), Brandon, Florida
  - Reliable Clinical Research, LLC (Site 100), Hialeah, Florida
  - A+ Research (Site 112), Miami, Florida
  - NextPhase Research Alliance at CANO HEALTH (Site 107), Miami, Florida
  - Ezy Medical Research (Site 106), Miami, Florida
  - Eminat LLC (Site 117), Plantation, Florida
  - Invictus Clinical Research Group, LLC (Site 101), Pompano Beach, Florida
  - Visionaries Clinical Research, LLC (Site 121), Atlanta, Georgia
  - Family Care Research (Site 114), Boise, Idaho
  - Cedar Crosse Research Center (Site 122), Chicago, Illinois
  - Massachusetts General Hospital (Site 110), Boston, Massachusetts
  - Oakland Medical Research Center (Site 108), Troy, Michigan
  - Cary Research Group (Site 111), Cary, North Carolina
  - Onsite Solutions (Site 118), Charlotte, North Carolina
  - STAT Research (Site 109), Springboro, Ohio
  - Toledo Institute of Clinical Research, Inc.(Site 105), Toledo, Ohio
  - Advanced Medical Trials (Site 104), Georgetown, Texas
  - Next Innovative Clinical Research (Site 115), Houston, Texas
  - Rio Grand Valley Clinical Research Institute (Site 120), Pharr, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed between November 09, 2020 to March, 30 2021. Subjects were recruited from ~25 sites across United States.
Period: Overall Study
Arm/Group | Camostat Mesilate | Placebo
Started | 194 | 101
Completed | 194 | 100
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat population includes all subjects who were randomized. [Note: Subjects may have more than one risk factor upon entry into study.]
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat Mesilate | Placebo | Total
Number analyzed (Participants) | 194 | 101 | 295
Age, Customized [Count of Participants; unit: Participants]
  < 55 years | 105 | 53 | 158
  > or = 55 years | 89 | 48 | 137
Sex: Female, Male [Count of Participants; unit: Participants] — The Intent-to-Treat population includes all subjects who were randomized.
  Participants
    Female | 108 | 61 | 169
    Male | 86 | 40 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 62 | 177
  Not Hispanic or Latino | 78 | 39 | 117
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 17 | 46
  White | 153 | 80 | 233
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression at Day 28
Description: Disease progression will be defined as the number of participants requiring hospitalization (including emergency room visit) or who die due to any cause within 28 days of randomization.
Time Frame: 28 days
Population: The Intent-to-Treat population includes all subjects who were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Participants | 10 | 6
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.787, Chi-squared — <0.05

2. Secondary Outcome: Survival Rate
Description: The overall survival rate (the number of randomized participants who survive up to Day 15 and Day 28).
Time Frame: Up to Day 15 and Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Participants
  Survival Status at Day 15 | 194 | 101
  Survival Status at Day 28 | 193 | 101

3. Secondary Outcome: Time to Fever Resolution
Description: Time (in days) from initiation of study treatment until normalization of fever (≤ 37.2 °C oral or tympanic) and sustained for at least 3 days only assessed in participants who experienced a fever within 1 day of enrollment up to Day 28.
Time Frame: Up to 28 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 18 | 5
Days | 3 [2.0 to 8.0] | 1 [1.0 to 1]

4. Secondary Outcome: Resolution of Viral Shedding
Description: Number of participants with no viral shedding (yes/no) using reverse transcriptase-polymerase chain reaction (RT-PCR) at Day 7, Day 15, and at early termination.
Time Frame: Day 1, Day 7 and Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Participants
  No Viral Shedding at Day 1 | 32 | 25
  No Viral Shedding at Day 7 | 77 | 36
  No Viral Shedding at Day 15 | 136 | 65

5. Secondary Outcome: Rate of Adverse Events and Serious Adverse Events
Description: Number of participants with Adverse events (AEs) and Serious adverse events (SAEs) of any grade from randomization up to Day 28.
Time Frame: 28 days
Population: A total of 295 subjects were randomized (2:1) to receive a 2-week course of Camostat (n=194) or placebo (n=101) One participant randomized to the placebo group decided to withdraw before taking the first dose of study drug, and one subject randomized to the placebo group was erroneously given Camostat mesilate (As Treated Population: Camostat mesilate, n=195 and placebo, n=99).
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 195 | 99
Participants
  Treatment Emergent Adverse Event (TEAE) | 17 | 13
  Serious TEAEs | 10 | 5

6. Secondary Outcome: Cumulative Rate of Grade 3 and 4 Adverse Events
Description: Cumulative number of participants with grade 3 and 4 AEs from randomization up to Day 28.
Time Frame: 28 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 195 | 99
Participants
  Grade 3 AEs | 6 | 0
  Grade 4 AEs | 1 | 1

7. Secondary Outcome: Rate of Discontinuation
Description: Number of participants that discontinued from study due to an AE/SAE (discontinued participants will be followed up to Day 28).
Time Frame: 28 days
Population: The Intent-to-Treat (ITT) population includes all subjects who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Participants | 11 | 5

8. Secondary Outcome: Laboratory Parameter - Platelet Count
Description: Clinical Laboratory Value of Platelet Count at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Population: The Intent-to Treat Population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
10^9 platelets/L
  Day 1 Platelet Count | 243 (71.69) | 252.1 (80.45)
  Day 15 Platelet Count | 288.3 (86.66) | 281.5 (83.22)

9. Secondary Outcome: Laboratory Parameter - Potassium Level
Description: Clinical laboratory value of Potassium Levels at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
mmol/L
  Day 1 Potassium Level | 4.26 (0.397) | 4.23 (0.391)
  Day 15 Potassium Level | 4.30 (0.363) | 4.29 (0.407)

10. Secondary Outcome: Laboratory Parameter - Aspartate Aminotransferase (AST)
Description: Clinical laboratory values of Aspartate Aminotransferase (AST) at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
U/L
  Day 1 AST | 24.6 (14.71) | 25.3 (12.33)
  Day 15 AST | 21.8 (10.18) | 21.8 (10.65)

11. Secondary Outcome: Laboratory Parameter - Alanine Aminotransferase (ALT)
Description: Clinical laboratory value of Alanine Aminotransferase (ALT) at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
U/L
  Day 1 ALT | 30.2 (27.58) | 29.0 (17.01)
  Day 15 ALT | 27.9 (20.1) | 27.9 (22.28)

12. Secondary Outcome: Laboratory Parameter - Alkaline Phosphatase (ALP)
Description: Clinical laboratory value of Alkaline Phosphatase (ALP) at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
U/L
  Day 1 ALP | 76.3 (24.44) | 80.5 (25.55)
  Day 15 ALP | 77.8 (27.60) | 78.6 (24.91)

13. Secondary Outcome: Laboratory Parameter - Gamma-Glutamyl Transferase (GGT)
Description: Clinical laboratory value of Gamma-Glutamyl Transferase (GGT) at Day 1 and Day 15
Time Frame: Day 1 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
U/L
  Day 1 GGT | 33.5 (25.61) | 33.4 (29.91)
  Day 15 GGT | 34.1 (30.50) | 31.1 (20.30)

14. Secondary Outcome: Vital Signs - Heart Rate
Description: Heart rate at Day 1, Day 7 and Day 15
Time Frame: Day 1, Day 7 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: Beats/Minute
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Beats/Minute
  Heart rate Day 1 | 81.2 (10.25) | 80.1 (10.48)
  Heart rate Day 7 | 81.2 (10.07) | 80.5 (9.09)
  Heart rate Day 15 | 79.8 (10.16) | 79.2 (9.94)

15. Secondary Outcome: Vital Signs - Blood Pressure
Description: Blood pressure (BP) at Day 1, Day 7 and Day 15
Time Frame: Day 1, Day 7 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
mmHg
  Systolic BP Day 1 | 128.7 (13.87) | 129.6 (13.97)
  Systolic BP Day 7 | 128.2 (16.61) | 129.2 (15.54)
  Systolic BP Day 15 | 128.1 (16.61) | 129.2 (15.54)
  Diastolic BP Day 1 | 80.7 (8.9) | 80.8 (7.43)
  Diastolic BP Day 7 | 80.2 (9.34) | 80.9 (9.6)
  Diastolic BP Day 15 | 78.9 (8.72) | 81.3 (10.65)

16. Secondary Outcome: Vital Signs - Peripheral Capillary Oxygen Saturation (SpO2)
Description: Peripheral Capillary Oxygen Saturation (SpO2) at Day 1, Day 7 and Day 15
Time Frame: Day 1, Day 7 and Day 15
Population: The Intent-to-Treat population includes all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: Percentage of SpO2
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 194 | 101
Percentage of SpO2
  SpO2 Day 1 | 97.3 (1.33) | 97.4 (1.3)
  SpO2 Day 7 | 97.3 (1.78) | 97.3 (1.43)
  SpO2 Day 15 | 97.6 (1.46) | 97.5 (2.22)

ADVERSE EVENTS:
Time Frame: 28 Days
Description: A total of 295 subjects were randomized (2:1) to receive a 2-week course of Camostat (n=194) or placebo (n=101) One participant randomized to the placebo group decided to withdraw before taking the first dose of study drug, and one subject randomized to the placebo group was erroneously given Camostat mesilate (As Treated Population: Camostat mesilate, n=195 and placebo, n=99).
Arm/Group | Camostat Mesilate | Placebo
All-Cause Mortality (participants affected / at risk) | 1/195 | 0/99
Serious Adverse Events (participants affected / at risk) | 10/195 | 5/99
Other Adverse Events (participants affected / at risk) | 8/195 | 9/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Camostat Mesilate (N=195) | Placebo (N=99)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2
Oxygen saturation decreased (Investigations) | 2 | 0
Delusion (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Camostat Mesilate (N=195) | Placebo (N=99)
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 1
Decreased apetite (Metabolism and nutrition disorders) | 1 | 0
Aguesia (Nervous system disorders) | 1 | 1
Anosmia (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04583592/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT04583592/SAP_001.pdf